CLINICAL TRIAL: NCT02035813
Title: DETECT IV - A Prospective, Multicenter, Open-label, Phase II Study in Patients With HER2-negative Metastatic Breast Cancer and Persisting HER2-negative Circulating Tumor Cells (CTCs).
Brief Title: DETECT IV - A Study in Patients With HER2-negative Metastatic Breast Cancer and Persisting HER2-negative Circulating Tumor Cells (CTCs).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prof. Wolfgang Janni (Other)
Responsible Party: Sponsor-Investigator, Prof. Wolfgang Janni, University hospital Ulm - Department of Gynecology, University of Ulm
Organization: University of Ulm (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D-IV; 2013-001269-18 (EudraCT Number)
Record Dates: First submitted 2014-01-12; First posted 2014-01-14 (Estimated); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: HER2-negative and Hormone-receptor Positive Metastatic Breast Cancer; HER2-negative Circulating Tumor Cells; Postmenopausal Female Patients
Keywords: metastatic breast cancer; circulating tumor cells; eribulin; ribociclib
MeSH Terms: conditions — Breast Neoplasms; Neoplastic Cells, Circulating | interventions — ribociclib; eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ribociclib in combination with standard endocrine therapy (Experimental): Postmenopausal female patients with hormone-receptor positive, HER2-negative metastatic breast cancer with HER2-negative circulating tumor cells (CTCs) and indication for standard endocrine therapy.
  Interventions: Drug: Ribociclib
- Eriubulin (Experimental): Patients with hormone-receptor positive, HER2-negative metastatic breast cancer and indication to chemother-apy or patients with triple-negative metastatic breast cancer, both with HER2-negative circulating tumor cells (CTCs).
  Interventions: Drug: Eribulin

INTERVENTIONS:
Drug: Ribociclib — Ribociclib/Everolimus in combination with endocrine therapy
  Other Names: Kisqali
  Arms: Ribociclib in combination with standard endocrine therapy
Drug: Eribulin
  Other Names: Halaven
  Arms: Eriubulin

SUMMARY:
Several studies have indicated that determining prevalence and number of circulating tumor cells (CTCs) at various time points during treatment may be an effective tool for assessing treatment efficacy in metastatic breast cancer (MBC). However, even if the prognostic value of CTCs in MBC is well understood, the role of both CTC prevalence and CTC phenotype in predicting treatment response needs further investigation. DETECT IV is a prospective, multicenter, open-label, phase II study in patients with HER2-negative metastatic breast cancer and persisting HER2-negative circulating tumor cells (CTCs). Additional research on CTC dynamics and characteristics will provide a better understanding of the prognostic and predictive value of CTCs and is one step into a more personalized therapy for MBC.

ELIGIBILITY:
Inclusion Criteria:

Both cohorts:

* Indication for an endocrine therapy (Histological confirmation of estrogen receptor positive (ER+) and/or progesterone receptor positive (PgR+) breast cancer).
* Up to two lines of previous cytostatic treatment for MBC.
* Any endocrine therapy in the history is allowed.
* Disease progression following prior treatment with endocrine therapy (endocrine therapy does not have to be the last therapy before inclusion in the trial).
* Postmenopausal women. The investigator must confirm postmenopausal status Postmenopausal status is defined either by

  * Age ≥ 55 years and one year or more of amenorrhea
* - Age < 55 years and one year or more of amenorrhea and postmenopausal levels of FSH and LH
* - Prior hysterectomy and has postmenopausal levels of FSH and LH
* - Surgical menopause with bilateral oophorectomy
* Everolimus cohort:
* Cholesterol ≤ 2.0 × ULN
* Ribociclib cohort:
* Standard 12-lead ECG values assessed by the local laboratory:
* - QTcF interval at screening < 450 msec (using Fridericia's correction)
* - Resting heart rate 50-90 bpm
* INR ≤ 1,5 (ribocilclib cohort)
* Patients must have the following laboratory values within normal limits or corrected to within normal lim-its with supplemets before the first dose of study medication:
* -Sodium
* -Potassium
* -Total calcium

For Eribulin only:

* Either hormone-receptor negative MBC or hormone-receptor positive MBC with indication for chemotherapy
* Up to three previous chemotherapy treatment lines for metastatic disease
* In case of patients of child bearing potential:

  * Negative pregnancy test (minimum sensitivity 25IU/L or equivalent units of HCG) within 7 days prior to recruitment
  * Contraception by means of a reliable method (i.e. non-hormonal contraception, IUD, a dou-ble barrier method, vasectomy of the sexual partner, complete sexual abstinence). Patient must consent in maintaining such contracep-tion until 3 months after completion of study treatment

Exclusion Criteria:

In General for both study cohorts:

1. Treatment with other investigational agents of any type or anticancer therapy during the trial, within 2 weeks prior to the start of treatment.
2. Adverse events due to prior anticancer therapy which are > Grade 1 (NCI CTCAE) and therapeutically relevant at time of treatment start.
3. Known HIV infection.
4. Current active hepatitis B or C, cliniclally relevant known liver dysfunction, e.g. according to Child Pugh Classifica-tion class B and C, or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gall-stones, liver metastases or stable chronic non-viral liver disease per investigator assessment).
5. Concurrent disease or condition that might interfere with adequate assessment or evaluation of study data, or any medical disorder that would make the patient's participation unreasonably hazardous.
6. Other malignant diseases within the last 3 years (apart from carcinoma in situ of the cervix or non-melanoma skin cancer)
7. Dementia, altered mental status, or any psychiatric or social condition which would prohibit the understanding or rendering of informed consent or which might interfere with the patient's adherence to the protocol.
8. Life expectancy < 3 months.
9. Male gender.

For Everolimus/Ribociclib only:

* Known hypersensitivity to any of the excipients of ribociclib, everolimus or any of the other given drugs.
* Known hypersensitivity to lecithin (soya) and pea-nuts (ribocilib-cohort)
* Disease or condition, which might restrain the ability to take or resorb oral medication. This includes malabsorption syndrome, requirement for intrave-nous (IV) alimentation, prior surgical procedures af-fecting absorption (for example resection of small bowel or stomach), uncontrolled inflammatory GI disease (e.g., Crohn's disease, ulcerative colitis) and any other diseases significantly affecting gas-trointestinal function as well as inability to swallow and retain oral medication for any other reason.

For Eribulin only:

* History of hypersensitivity reactions attributed to eribulin.
* Pre-existing neuropathy grade 3 or higher.
* Severe Congenital long QT syndrome.
* Pregnancy or nursing.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 8-12 weeks
  Time interval from randomization until progressive disease (PD) or death from any cause, whichever comes first

SECONDARY OUTCOMES:
Overall response rate | 8-12 weeks
  Rate of complete (CR) and partial responses (PR) in patients with whom target lesions were defined
Disease control rate (DCR) | 8-12 weeks
  rate of patients who were assessed as having a PR or a CR or who had stable disease (SD) for at least 6 months
Overall survival (OS) | 4 weeks
  Time from randomization until death of any cause
Dynamic of CTCs | 8-12 weeks
  Descriptive statistics of regular CTC counts
For Everolimus/Ribociclib cohort only: Levels of pS6 | 8-12 weeks
  Descriptive statistics of pS6 levels at baseline, at first radiological tumor assessment after about 12 weeks, and at the time of progression
For Everolimus/Ribociclib cohort only: Change in the activation of the PI3K/Akt/mTOR-pathway in CTCs | 8-12 weeks
  Descriptive statistics of changes in the activation of the PI3K/Akt/mTOR-pathway in CTCs as assessed by longitudinal comparisons (at baseline, after 12 weeks, at time of progression)
For Everolimus/Ribociclib cohort only: Estrogen-receptor 1 (ESR-1) mutations in CTCs | 8-12 weeks
  Estrogen-receptor 1 (ESR-1) mutations in CTCs at baseline, after 12 weeks and at time of progression
For Eribulin cohort only: New metastasis-free survival (nMFS) | 8-12 weeks
  New metastasis-free survival (nMFS), defined as time from recruitment to death or progression due to appearance of a new metastasis, whichever comes first. If a patient has not had an event, nMFS is censored at the date of last adequate tumor as-sessment

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Fehm, MD, PhD, Principal Investigator — University Hospital Düsseldorf -Department of Gynecology; Wolfgang Janni, MD, PhD, Study Director — University Hospital Ulm -Department of Gynecology
Locations (1):
- University Hospital Ulm -Department of Gynecology, Ulm, Baden-Wurttemberg, Germany

REFERENCES:
- See also: Related Info — http://www.detect-studien.de